CLINICAL TRIAL: NCT06640972
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of RDX-002 on Postprandial Triglycerides in Patients Discontinuing the Glucagon-like Peptide-1 (GLP-1) Agonists, Semaglutide or Tirzepatide, for the Treatment of Obesity
Brief Title: Effects of RDX-002 on Postprandial Triglycerides in Patients Discontinuing GLP-1 Agonists
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RDX-002-024-011
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Triglycerides; Weight Gain Trajectory; Cholesterol, Elevated
Keywords: RDX-002; GLP1; triglyceride; obesity; semaglutide; tirzepatide; microsomal triglyceride transfer protein inhibitor; MTP
MeSH Terms: conditions — Body-Weight Trajectory; Hypercholesterolemia; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational drug (Experimental): The effect of 12 weeks of treatment with RDX-002 on postprandial TGs, fasting levels of cholesterol, and body weight among patients who have recently discontinued treatment with the GLP-1 agonists, semaglutide or tirzepatide, for obesity.
  Interventions: Drug: RDX-002
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDX-002 — Gut-specific microsomal triglyceride transfer protein (MTP) inhibitor
  Arms: Investigational drug
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug RDX-002 works to treat high levels of fat (known as triglycerides, or TGs) in the blood in adults. It will also learn about the safety of drug RDX-002. The main question it aims to answer is if treatment with RDX-002 will lower triglycerides after a high-fat meal in patients who have recently stopped treatment with semaglutide or tirzepatide for obesity. The trial will also examine the effect of RDX-002 on body weight and fasting levels of cholesterol.

Researchers will compare RDX-002 to a placebo (a look-alike substance that contains no drug) to see if RDX-002 works to reduce triglycerides.

Participants will:

Take drug RDX-002 or a placebo every day for 12 weeks Visit the clinic once every 4 weeks for checkups and tests

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group study that will be conducted at a single study site in the United States (US).

Patients who have planned discontinuation of semaglutide or tirzepatide treatment for obesity, have lost ≥10% or 10 Killigrams (kg) of their original body weight and are aged 18 to 65 years will be eligible for Screening. The study will assess the efficacy of 12 weeks of treatment with 200 mg twice daily (BID) RDX-002 or placebo on the mean percentage change from baseline on postprandial TGs among patients who have recently discontinued treatment with semaglutide or tirzepatide for obesity. The trial will also examine the impact of RDX-002 on body weight and fasting levels of cholesterol.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to the conduct of any study specific procedures;
2. Planned or willing discontinuation of semaglutide or tirzepatide for the treatment of obesity prior to randomization (Visit T1/Day 1) through the end of study (EOS);
3. Lost ≥10% or 10 kg of original (pre-GLP-1 baseline) body weight with semaglutide or tirzepatide;
4. Males and females aged 18 to 65 years (both inclusive) at Screening (Visit S1);
5. A hemoglobin A1C (HbA1c) of <6.5% at Screening (Visit S1);
6. A 12-lead (electrocardiograph) ECG at Screening (Visit S1) which, in the opinion of the investigator, had no abnormalities that compromised safety in this study;
7. Males and nonpregnant, nonlactating females. Females must be either of non-childbearing potential or use appropriate birth control methods and have a negative pregnancy test at Screening

Exclusion Criteria:

1. Type 1 or Type 2 diabetes;
2. Recent (within 3 months prior to the Screening visit [Visit S1]) cardiovascular event or planned or recent cardiovascular surgery or intervention. Patients with implantable pacemakers or automatic implantable cardioverter defibrillators may be considered if deemed by the investigator to be stable for the previous 3 months;
3. Uncontrolled hypertension, defined as systolic blood pressure (SBP) >160 mmHg and diastolic blood pressure (DBP) >100 millimeters of mercury (mmHg) after being in supine position for 5 minutes;
4. Total fasting (minimum of 10 hours) TGs ≥400 milligrams per deciliter (mg/dL) (4.5 millimoles per liter (mmol/L)) at Screening (Visit S1);
5. Fasting glucose >126 mg/dL at Screening (Visit S1);
6. Uncontrolled hypothyroidism, including thyroid stimulating hormone (TSH) >1.5 × the upper limit of normal (ULN) at Screening (Visit S1); patients stabilized on thyroid replacement therapy for at least 6 weeks prior to randomization (Visit T1/Day 1) are allowed; Liver disease or dysfunction, including positive serology or hepatitis B and/or C or significant elevations in certain liver function tests
7. Renal dysfunction or glomerulonephritis, including estimated glomerular filtration rate (eGFR; using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] 2021 formula) <60 milliliters per minute (mL/min) at Screening (Visit S1).
8. Gastrointestinal conditions or procedures (including weight loss surgery; e.g., Lap-Band® or gastric bypass) except uncomplicated cholecystectomy and appendectomy that may affect drug absorption;
9. Known history of hematologic or coagulation disorders or a hemoglobin level <10.0 grams/deciliter (g/dL) at Screening (Visit S1);
10. Active malignancy, including those requiring surgery, chemotherapy, and/or radiation in the past 5 years. Nonmetastatic basal or squamous cell carcinoma of the skin and cervical carcinoma in situ are allowed;
11. Unexplained creatine kinase (CK) >3 × ULN at any time prior to randomization (i.e., not associated with recent trauma or physically strenuous activity). Patients with an explained CK elevation must have single repeat CK ≤3 × ULN prior to randomization;
12. History of drug or alcohol abuse within the last 2 years or reported current consumption of >14 alcoholic drinks/week, or any illicit drug use (checked positive for standard drug screening panel). Patients testing positive for tetrahydrocannabinol (THC) (whether prescribed or not) and for amphetamine derivatives prescribed by and under the care of a health care practitioner (except for weight management) can be enrolled after evaluation and at the discretion of the investigator;
13. Inability to follow the required minimum 2 meals a day, or unwillingness to consume meal on both study test occasions, or inability to fast, as required during the study;
14. Blood donation, participation in multiple blood draws, clinical study, major trauma, blood transfusion or surgery with or without blood loss within 30 days prior to randomization (Visit T1/Day 1);
15. Use of any experimental or investigational drugs except GLP-1 agonists within 30 days or 5 half-lives (whichever is longer) prior to Screening (Visit S1);
16. Use of any prohibited diabetes or other weight loss drugs prior to or during the study (as specified) unless meeting specific rescue criteria:
17. Recent (within 30 days unless otherwise specified) initiation or discontinuation of lipid-lowering medications. Consistent background use is allowed;
18. An employee or contractor of the facility conducting the study, or a family member of the principal investigator, co-investigator, or any Sponsor personnel;
19. Pregnant, breastfeeding, or intending to become pregnant within 30 days after study completion or last dose of study drug;
20. A medical or situational (i.e., geographical) finding that, in the investigator's opinion, may compromise the patient's safety or ability to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 12 weeks
  Difference in the mean percent change in the incremental postprandial TG area under the curve (AUC) in patients treated with RDX 002 as compared with placebo at Week 12.

SECONDARY OUTCOMES:
Change in mean percent body weight | 12 weeks
  Difference in the mean percent change from baseline in body weight in patients treated with RDX-002 as compared with placebo at Week 12.
LDL-C | 12 weeks
  Difference in the mean percent change from baseline in LDL-C in patients treated with RDX-002 as compared with placebo at week 12.
Change in body weight by 5% | 12 Weeks
  Difference in the proportion of patients treated with RDX-002 exhibiting at least a 5% increase from baseline in body weight as compared with placebo at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Stamp, PhD, PA-C, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Saint Paul, Minnesota, United States